CLINICAL TRIAL: NCT07071623
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy and Safety of MK-8527 Oral Once-Monthly as HIV-1 Preexposure Prophylaxis in Women
Brief Title: A Study of MK-8527 to Prevent Human Immunodeficiency Virus Type 1 (HIV-1) (MK-8527-010)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8527-010; MK-8527-010 (Other: MSD)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Pre-Exposure Prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-8527 + Placebo to FTC/TDF (Experimental): Participants will receive 11 mg MK-8527 once monthly (QM) and placebo matched to Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) once daily (QD) for up to approximately 2 years. Participants will then receive open-label 200 mg FTC/245 mg TDF QD for an additional 28 days.
  Interventions: Drug: MK-8527; Drug: Placebo matched to FTC/TDF
- FTC/TDF + Placebo to MK-8527 (Active Comparator): Participants will receive 200 mg FTC/245 mg TDF QD and placebo matched to MK-8527 QM for up to approximately 2 years. Participants will then receive open-label 200 mg FTC/245 mg TDF QD for an additional 28 days.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil (FTC/TDF); Drug: Placebo matched to MK-8527

INTERVENTIONS:
Drug: MK-8527 — Oral tablet
  Arms: MK-8527 + Placebo to FTC/TDF
Drug: Emtricitabine/tenofovir disoproxil (FTC/TDF) — Oral tablet
  Other Names: Truvada; Emtricitabine/Tenofovir Disoproxil Fumarate
  Arms: FTC/TDF + Placebo to MK-8527
Drug: Placebo matched to MK-8527 — Placebo oral tablet matched to MK-8527
  Arms: FTC/TDF + Placebo to MK-8527
Drug: Placebo matched to FTC/TDF — Placebo oral tablet matched to FTC/TDF
  Arms: MK-8527 + Placebo to FTC/TDF

SUMMARY:
Researchers are looking for new medicines to prevent HIV-1 (Human Immunodeficiency Virus Type 1) infection.

The goals of this study are to learn:

* If taking MK-8527 once a month works to prevent HIV-1 infection better than a standard (usual) pre-exposure prophylaxis (PrEP) taken once a day
* About the safety of MK-8527 and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is confirmed Human Immunodeficiency Virus (HIV)-uninfected based on negative HIV-1/HIV-2 test results
* Has been sexually active (2 vaginal intercourse encounters with cisgender male individual(s) within the last 3 months)
* Was assigned female sex at birth and is cisgender.
* Weighs ≥35 kg

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has hypersensitivity or other contraindication to any component of the study interventions
* Has evidence of acute or chronic hepatitis B infection
* Has a history of malignancy within 5 years of screening except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Has taken cabotegravir, lenacapavir, or any other long-acting HIV prevention product at any time
* Is receiving or is anticipated to require any prohibited therapies from 30 days prior to Day 1 through the study duration
* Has received an HIV vaccine at any time (ie, through past participation in an investigational clinical study) or monoclonal antibodies to HIV within 12 months before Day 1

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must be assigned female sex at birth and cisgender.
Enrollment: 4580 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adjudicated Human Immunodeficiency Virus Type 1 (HIV-1) Infection | Up to ~2 years
  The number of participants with adjudicated HIV-1 infection will be presented.
Number of Participants who Experience At Least One Adverse Event (AE) | Up to ~2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experienced AEs will be presented.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to ~2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that discontinued study intervention due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- Kenya (4):
  - UW - KNH; Rachuonyo County Hospital ( Site 0006), Homabay County, Homa Bay County
  - Partners in Health and Research Development (PHRD) ( Site 0002), Thika, Kiambu County
  - KEMRI-CMR-RCTP ( Site 0003), Nairobi, Kisumu County
  - Kargeno Research & Policy Hub ( Site 0007), Kisumu
- South Africa (21):
  - Synergy Biomed Research Institute ( Site 0040), East London, Eastern Cape
  - Foundation For Professional Development ( Site 0031), Ndevana, Eastern Cape
  - Josha Research ( Site 0045), Bloemfontein, Free State
  - Wits RHI Ward 21 Clinical Research site ( Site 0022), Johannesburg, Gauteng
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 0048), Johannesburg, Gauteng
  - Perinatal HIV Research Unit (PHRU) ( Site 0033), Johnnesburg, Gauteng
  - Setshaba Research Centre ( Site 0032), Pretoria, Gauteng
  - SA Medical Research Council - Chatsworth Clinical Research Site ( Site 0026), Chatsworth, KwaZulu-Natal
  - SA Medical Research Council - Botha's Hill Clinical Research Site ( Site 0035), Durban, KwaZulu-Natal
  - CAPRISA eThekwini Clinical Research Site ( Site 0030), Durban, KwaZulu-Natal
  - Wits Maternal Adolescent and Child Health Research Unit (WMRU) ( Site 0027), Durban, KwaZulu-Natal
  - Umlazi Clinical Research Site ( Site 0047), Durban, KwaZulu-Natal
  - SYNAPSE Research Clinic ( Site 0043), Edendale, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic ( Site 0028), Ladysmith, KwaZulu-Natal
  - SA Medical Research Council - Phoenix Clinical Research Site ( Site 0037), Phoenix, KwaZulu-Natal
  - CAPRISA Vulindlela Clinical Research Site ( Site 0029), Pietermaritzburg, KwaZulu-Natal
  - Africa Health Research Institute (AHRI) - Mtubatuba ( Site 0049), Somkhele - Mtubatuba, KwaZulu-Natal
  - SA Medical Research Council - Verulam Clinical Research Site ( Site 0036), Verulam, KwaZulu-Natal
  - Desmond Tutu Health Foundation. Philippi Village ( Site 0024), Cape Town, Western Cape
  - DTHF Masiphumelele Clinical Research Site ( Site 0023), Cape Town, Western Cape
  - Vuka Research Clinic ( Site 0025), Khayelitsha, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com